CLINICAL TRIAL: NCT03268876
Title: The INFLUENCE of Cytoreduction on Patient Reported Outcomes in Patients With Epithelial Ovarian Cancer
Brief Title: The INFLUENCE of Cytoreduction on PRO in EOC
Acronym: INFLUENCE
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/941
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial ovarian cancer; Surgery; Quality of life
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and tumor biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epithelial ovarial cancer: Patients primary treated with primary surgery for advanced epithelial ovarian cancer (> stage IIa) at the participating institutions will be asked to participate.

SUMMARY:
Based on an improved understanding of how the extent of successful cytoreduction is influenced both by inherent tumor biological characteristics as well as the aggressiveness of the surgical approach this project aims to better define the value of cytoreduction and to use the knowledge gained to develop more individualized therapy and follow-up. This will be achieved through a translational biomedical research approach. Due to the research group's traditions clinical phenotyping, biomarker identification, and clinical trials will be the focus.

DETAILED DESCRIPTION:
The patients will be recruited at their follow-up appointment after their surgery. At this consultation the patient will be informed about the final diagnosis and extent of disease and a plan for their further chemotherapeutic treatment will be developed. All patients will be offered carboplatin AUC 5 and paclitaxel 175mg/m2 q3w for 6 cycles [+ bevacizumab 7.5mg/kg q3w for 18 cycles in high-risk women of recurrence (IIIc not maximal debulked with a rest tumor of >1 cm2 and stage IV)]. In they fulfill the inclusion criteria and agree the inform consent formula will be signed. During the screening period the study team will secure that the necessary information needed is available and study specific test and analysis will be undertaken. After inclusion the study specific consultations will be scheduled coinciding with the patient regular appointments for treatment and follow-up. The patients will be followed at predetermined time points (after finalizing the chemotherapy; and every 3 months thereafter for 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer
* Stage > II
* ECOG < II
* Treated with primary surgery followed by chemotherapy
* Willing to participate and to sign the informed consent

Exclusion Criteria:

* < 18 years old
* Borderline and non-epithelial ovarian tumors
* Stage < II
* Advanced ovarian cancer submitted to neoadjuvant chemotherapy
* ECOG 3-4
* Pregnancy
* Severe cardiopulmonary disease
* Patients participating in QoL intervention studies

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients primary treated with primary surgery for advanced epithelial ovarian cancer at the participating institutions will be asked to participate.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Global Health Score | 2 years
  Is there a relationship between QOL score and immunologic profiling in biological samples?

CONTACTS AND LOCATIONS:
Overall Officials: Line Bjørge, MD, PhD, MBA, Principal Investigator — Helse-Bergen HF
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Sørlandet sykehus HF, Kristiansand
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: Undecided